CLINICAL TRIAL: NCT00721994
Title: Cormet Resurfacing Hip System Post PMA Approval Study (PMA #P050016)Pre-market (IDE) Study Group 10 Year Follow-Up With Metal Ion and Renal Function Data Collection Clinical Investigation Plan
Brief Title: Post-PMA Approval Study: 10 Year Follow-Up IDE Subjects
Acronym: PAS:IDE
Status: Completed | Type: Observational
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: PAS: IDE subjects
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis
Keywords: hip resurfacing; osteoarthritis; avascular necrosis; rheumatoid arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood specimens for metal ion testing and renal function testing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: IDE subjects who received the Cormet Hip Resurfacing device
  Interventions: Device: Cormet Hip Resurfacing System

INTERVENTIONS:
Device: Cormet Hip Resurfacing System — Cormet Hip Resurfacing System
  Other Names: Corin Cormet

SUMMARY:
primary endpoint of this Study is maintenance of "at least good clinical status" for a period of 10 years following initial implantation among Cormet procedures enrolled inthe pre-market IDE.

DETAILED DESCRIPTION:
Maintaining "at least good clinical status" will be determined based upon the composite clinical success (CCS) criterion which includes no revision, removal, or replacement of any device component and a Harris Hip Total score of greater or equal to 80 points.

ELIGIBILITY:
Inclusion Criteria:

* subjects enrolled in the Cormet IDE study at the 5 identified clinical sites
* Individuals who agree to participate in the study by signing the informed patient consent form

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IDE study subjects at 5 IDE study sites
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2008-05; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
to monitor the clinical performance of the Cormet implant system for a period of up to 10 years postoperative in order to confirm that there are no unexpected reductions in device performance following PMA approval | 10 years

SECONDARY OUTCOMES:
Harris Hip Score components including total score, pain, function and range of motion | 10 years
device survival | 10 years
device related adverse events | 10 years
radiographic evaluation including radiolucencies, component migration, and femoral subsidence and tilt | 10 years
whole blood trace metals and renal function | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Trier, Ph.D., Study Director — Corin
Locations (5):
- United States (5):
  - Space Coast Orthopaedics Ctr., Merritt Island, Florida
  - Kennedy White Orthopedics, Sarasota, Florida
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Good Samaritan Hospital, Baltimore, Maryland
  - Cleveland Center for Joint Reconstruction, Cleveland, Ohio